CLINICAL TRIAL: NCT03628118
Title: A Research on Hidden Blood Loss in Open Radical Hysterectomy and Pelvic Lymphadenectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2018-07-130
Record Dates: First submitted 2018-08-05; First posted 2018-08-14 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hidden Blood Loss; Open Radical Hysterectomy; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- open radical hysterectomy: The patients who would undergo "open radical hysterectomy" procedure.

SUMMARY:
The aim of this cross-sectional study is to evaluate the hidden blood loss in patients who underwent open radical hysterectomy and identity its risk factors.

DETAILED DESCRIPTION:
The electronic medical data of 100 patients who undergo open radial hysterectomy in the following year to treat cervical cancer will be analyzed retrospectively in this study. The amount of hidden blood loss will be calculated according to Gross's formula. And multiple linear regression analysis will be employed to identify its risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. Females aged 20-80 who are confirmed with cervical cancer and are treated with open radical hysterectomy and pelvic lymphadenectomy.

Exclusion Criteria:

1. Pregnancy, lactation, postmenopause, or planned pregnancy within two years;
2. Suspected or identified as other tumors of genital tract;
3. History of hyperparathyroidism, infectious diseases (tuberculosis, AIDS), autoimmune diseases, or digestive system diseases (malabsorption, crohn disease and dysentery);
4. Other diseases or heavy injuries that will interfere with the results;
5. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned sample size was based on data from a previous study, in which the standard deviation was 5. We assumed an one-tailed α error of 0.05 and a sampling error of 1.0. we propose to enroll 105 participants and allow for a dropout rate of 10% for an effective sample size of 100.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
the volume of hidden blood loss (mL) | 10 months after surgery
  the volume of invisible blood loss occurring in patients who undergo open radical hysterectomy applying Gross's formula

SECONDARY OUTCOMES:
the risk factors of hidden blood loss | 10 months after surgery
  Performing multiple linear regression analysis with SPSS 17.0, we plan to identify the factors which may increase the volume of hidden blood loss from possible factors like hypertension, diebetes, etc.
the volume of total blood loss (mL) | 10 months after surgery
  the vomule of patients' blood loss through the whole perioperative time according to the method of Nadler
the volume of visible blood loss (mL) | 10 months after surgery
  the visible blood loss including the blood in the suction bottle and in weighed compresses during the operation and the drainage volume after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- TING LI, Wenzhou, Zhejiang, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03628118/Prot_SAP_000.pdf